CLINICAL TRIAL: NCT01049243
Title: An Open-Label Study Evaluating the Efficacy of Fluocinonide Cream 0.1% (Vanos) in Subjects With Atopic Dermatitis
Brief Title: A Study Evaluating the Efficacy of Fluocinonide Cream 0.1% (Vanos) in Subjects With Atopic Dermatitis
Acronym: Vanos
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006468
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Open-Label; Topical; Cream; Eczema; Vanos
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Fluocinonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluocinonide Cream 0.1% (Other): Fluocinonide Cream 0.1% open label
  Interventions: Drug: Fluocinonide Cream 0.1%

INTERVENTIONS:
Drug: Fluocinonide Cream 0.1% — 0.1% Cream, One Application, Twice Daily, 14 Days
  Other Names: Vanos

SUMMARY:
The purpose of this research study is to better understand how fluocinonide cream 0.1% (Vanos®) works when people use it to treat atopic dermatitis for just a few days.

DETAILED DESCRIPTION:
This is a single center study. This is an open label study of fluocinonide cream 0.1% (Vanos™) for subjects with mild to severe atopic dermatitis with an assessment of 2 to 4 on the Investigator Global Assessment scale (Appendix B). Up to 20 subjects age 12 and above will be enrolled after providing informed consent. All subjects will receive the study medication, fluocinonide cream 0.1% (Vanos™). Each subject will be instructed to use fluocinonide cream 0.1% (Vanos™) twice daily for three consecutive days (for a total of 6 doses). The study period will last for approximately 2 weeks. Subjects will be evaluated at baseline and Day 2 or 3 (as needed to achieve 6 doses), day 7 and day 14 (or end of study). Subjects will not apply any study drug after the 6 doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with mild to severe atopic dermatitis, 12 years of age or older, that agree to participate and provide written consent (and assent if applicable)
* Have an Investigator Global Assessment of mild to severe atopic dermatitis (IGA rating of 2 - 4 in the Investigator Global Assessment (Appendix B))
* Percentage of overall body surface are of involvement (BSA) must be ≥2%
* Women of child bearing potential will be allowed to participate in the study, and these subjects will be required to use at least one form of birth control

Exclusion Criteria:

* Use within 4 weeks of baseline of systemic anti-inflammatory medication, which may influence study outcome, such as systemic corticosteroids
* Application or use within 2 weeks of baseline of topical corticosteroid medications or topical anti-inflammatory medication, which may influence study outcome
* Presence of a concurrent medical condition, which is determined by the investigator to potentially interfere with study outcomes or patient assessments
* Introduction of any other prescription medication, topical or systemic, for atopic dermatitis while participating in the study
* Amount of disease involvement that would require >60 gm of cream in a 1 week period
* Subjects with known allergy or sensitivity to topical Vanos™ cream or components
* Pregnant women and women who are breastfeeding are to be excluded. Women of childbearing potential will be allowed to participate in the study, and these subjects will be required to use at least one form of birth control.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from IRB approved advertising and the Wake Forest University Health Sciences Dermatology Clininc
Groups:
- Vanos: Single group; 0.1% Cream, One Application, Twice Daily, 14 Days
Period: Overall Study
Arm/Group | Vanos
Started | 20
Completed | 18
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Group
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 27 [17 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Investigator Global Assessment of Atopic Dermatitis Severity From Baseline to Day 2/3.
Description: Use of the Investigator's Global Assessment (IGA) score, a subjective scale measuring disease severity. Based on a 6-point scale from 0 (completely clear) to 5 (very severe). Defined score of 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe.
Time Frame: Baseline to 3 days
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 20
Scores on a scale | -0.72 (0.57)

2. Secondary Outcome: Change in Investigator Global Assessment of Atopic Dermatitis Severity From Baseline to Day 14.
Description: as for outcome 1
Time Frame: Baseline to 14 days
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Fluocinonide Cream 0.1%
Number analyzed (Participants) | 20
units on a scale | 2.4 [1.7 to 3.2]

ADVERSE EVENTS:
Arm/Group | Single Group
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No